CLINICAL TRIAL: NCT04331015
Title: Positive Predictive Value of Machine Learning Tools (Audiogene v4.0) for Diagnosing DFNA9 in a Large Series of p.Pro51Ser Variant Carriers in COCH.
Brief Title: Artificial Intelligence in Diagnosis of DFNA9
Acronym: DFNA9
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JessaH-5-ORL
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: DFNA9; Sensorineural Hearing Loss
Keywords: COCH; DFNA9; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Audiometry, Pure-Tone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pure tone audiometry — pure tone audiometry

SUMMARY:
To study the positive predictive value of Audiogene v.4.0 open source online machine learning tool in accurately predicting DFNA9 (DeaFNess autosomal dominant ninth) as top 3 gene loci in a large series of genetically confirmed c.151C>T,p.Pro51Ser (p.P51S) variant carriers in COCH (coagulation factor C Homology).

DETAILED DESCRIPTION:
DFNA9 is an autosomal dominant hereditary adult-onset and progressive sensorineural hearing loss which is associated wit vestibular deterioration.

Today, artificial intelligence plays an increasing role in diagnosis of Mendelian hearing losses and in fitting of cochlear implants. An application of this kind is the open source program, Audiogene v4.0, which was elaborated by the Center for Bioinformatics and Computational Biology, University of Iowa City, Iowa, USA. The shape of the audiogram (audioprofile) is easily recognizable in many autosomal dominantly inherited hearing losses. Machine learning based software tools, such as Audiogene v4.0, which was originally developed for prioritizing loci for the Sanger sequencing, could help the clinicians in early diagnosis of DFNA9. This tool only need subjects' age and hearing thresholds (decibel hearing loss (dB HL)) at frequency range of 0.125 - 8 kHz (kiloHerz), left, right or binaural average in order to predict top 3 gene loci according to the data entered in the program.

Goal: to use auditory data of a large series of genetically confirmed p.P51S variant carriers causing DFNA9, which were previously collected for the genotype-phenotype correlation study which terminated recently.

All individual left and right sided hearing thresholds (ranging from 0.125 to 8kHz, with the exception of 1.5 kHz) as well as binaural averaged thresholds were run through Audiogene v4.0.

Descriptive statistics were assessed and statistical analysis was carried out to check for possible differences between age or hearing thresholds between the carrier group with accurate prediction against the carrier group with inaccurate prediction.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* genetically confirmed c.151 C>T, p.Pro51Ser variant carrier in COCH gene
* not contra-indication for audiometric testing

Exclusion Criteria:

* <18 years
* no carrier status for c.151C>T, p.Pro51Ser
* no auditory data available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A large cohort of 111 genetically confirmed p.P51S variant carriers, of whom audiometric data was collected from
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
hearing threshold | 1 hour
  audiometry (pure tone) decibel hearing level (dB HL) left, right ear , binaural average
age | 1 hour
  years, age at time of audiometry
prediction gene locus | 1 hour
  top 3 gene loci as predicted by Audiogene v4.0 machine learning tool

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Van Rompaey, MD,PhD, Study Director — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - Jessa Hospital, Hasselt, Limburg
  - University of Antwerp, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taylor KR, Deluca AP, Shearer AE, Hildebrand MS, Black-Ziegelbein EA, Anand VN, Sloan CM, Eppsteiner RW, Scheetz TE, Huygen PL, Smith RJ, Braun TA, Casavant TL. AudioGene: predicting hearing loss genotypes from phenotypes to guide genetic screening. Hum Mutat. 2013 Apr;34(4):539-45. doi: 10.1002/humu.22268. Epub 2013 Feb 19. PMID 23280582
- See also: audiogene v4.0 — http://audiogene.eng.uiowa.edu/